CLINICAL TRIAL: NCT00843856
Title: Mycophenolate Mofetil and Tacrolimus vs Tacrolimus Alone for the Treatment of Idiopathic Membranous Glomerulonephritis (IMG)
Brief Title: Mycophenolate Mofetil and Tacrolimus Versus Tacrolimus for the Treatment of Idiopathic Membranous Glomerulonephritis
Acronym: MTAC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13HH1282; 2008-001009-41 (EudraCT Number)
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Results first posted 2019-12-12 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-11

CONDITIONS: Glomerulonephritis, Membranous
Keywords: Glomerulonephritis
MeSH Terms: conditions — Glomerulonephritis, Membranous; Glomerulonephritis | interventions — Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tacrolimus (Active Comparator): Intervention type -drug tacrolimus therapy 2mg bd adjust to obtain levels of 5-12ng/L
  Interventions: Drug: tacrolimus
- tacrolimus and mycophenolate mofetil (Active Comparator): tacrolimus 2mgs bd (adjusted to obtain levels 5-12mg/L and mycophenolate mofetil 500mg bd adjusted to obtain levels 1.5-3mg/L
  Interventions: Drug: tacrolimus and mycophenolate mofetil

INTERVENTIONS:
Drug: tacrolimus — tacrolimus 2mgs bd adjusted to obtain levels of 5-12ng/ml
  Other Names: prograff
  Arms: tacrolimus
Drug: tacrolimus and mycophenolate mofetil — tacrolimus 2mg bd adjusted to achieve levels of 5-12ng/L mycophenolate mofetil 500mgs bd adjusted to achieve levels of 1.5-3mg/L
  Other Names: prograf; cellcept
  Arms: tacrolimus and mycophenolate mofetil

SUMMARY:
Study Hypothesis: When mycophenolate mofetil is added to tacrolimus in the treatment of membranous glomerulonephritis it is likely to improve the initial response to treatment and reduce the risk of relapse on stopping therapy.

DETAILED DESCRIPTION:
Membranous nephropathy is a common cause of nephrotic syndrome in adults. It is difficult to treat and if persistent leads to end stage renal failure in a significant number of patients. It is currently treated in this institution with tacrolimus monotherapy. This is effective in the majority of patients in reducing proteinuria but the remissions are often partial and patients tend to relapse when the tacrolimus treatment is stopped. We propose to use mycophenolate mofetil in combination with tacrolimus with the aim of obtaining a more complete initial response to treatment, a decreased rate of relapse on withdrawal of therapy and less progression of renal failure. This will be a randomised control trial, patients will be randomised to receive treatment with tacrolimus alone (our current standard therapy)or treatment with tacrolimus and mycophenolate mofetil. Participants will receive treatment for up to 2 years and then be monitored for relapse of their nephrotic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic membranous glomerulonephritis on renal biopsy
* Proteinuria - protein/creatinine ratio (PCR) > 100 units with hypoalbuminaemia or PCR > 300 units with normal serum albumin despite 3 months treatment with maximum tolerated doses of ace inhibitors and angiotensin 2 antagonists (or shorter if life threatening complications of nephrotic syndrome require institution of immediate immunosuppression)
* Male or female patients aged 18 to 80 years

Exclusion Criteria:

* Hepatitis B hepatitis C or HIV positive
* Malignancy (all patients must have a CT chest abdomen and pelvis and other investigations if clinically indicated)
* Untreated infection
* Females who are pregnant, breast feeding, or at risk of pregnancy and not using a medically acceptable form of contraception
* Any condition judged by the investigator that would cause the study to be detrimental to the patient

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-03-03 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan Griffith, MBChB PhD, Principal Investigator — Imperial College London
Locations (1):
- Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nikolopoulou A, Condon M, Turner-Stokes T, Cook HT, Duncan N, Galliford JW, Levy JB, Lightstone L, Pusey CD, Roufosse C, Cairns TD, Griffith ME. Mycophenolate mofetil and tacrolimus versus tacrolimus alone for the treatment of idiopathic membranous glomerulonephritis: a randomised controlled trial. BMC Nephrol. 2019 Sep 6;20(1):352. doi: 10.1186/s12882-019-1539-z. PMID 31492152
- [Derived] von Groote TC, Williams G, Au EH, Chen Y, Mathew AT, Hodson EM, Tunnicliffe DJ. Immunosuppressive treatment for primary membranous nephropathy in adults with nephrotic syndrome. Cochrane Database Syst Rev. 2021 Nov 15;11(11):CD004293. doi: 10.1002/14651858.CD004293.pub4. PMID 34778952

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tacrolimus | Tacrolimus and Mycophenolate Mofetil
Started | 20 | 20
Completed | 19 | 18
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tacrolimus | Tacrolimus and Mycophenolate Mofetil | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Median (Full Range); unit: years] | 55 [24 to 68] | 48 [28 to 66] | 51 [24 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 11 | 13 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 20 | 20 | 40
Serum albumin [Median (Full Range); unit: g/L] | 17 [8 to 30] | 18 [11 to 27] | 17.5 [8 to 30]
Estimated glomerus filtration rate (GRF) [Median (Full Range); unit: mls/min/1.73m^2] | 109 [44 to 142] | 121 [63 to 201] | 115 [44 to 201]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patient Who Gained Remission From the Nephrotic Syndrome
Description: Efficacy of mycophenolate in preventing relapse of nephrotic syndrome secondary to membranous glomerulonephritis on withdrawal of tacrolimus therapy.
Time Frame: 10-109 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Tacrolimus | Tacrolimus and Mycophenolate Mofetil
Number analyzed (Participants) | 16 | 19
Participants | 8 | 8
Statistical Analysis 1: Comparison: Tacrolimus vs Tacrolimus and Mycophenolate Mofetil; Test type: Superiority; p = 0.7, Fisher Exact

2. Secondary Outcome: Number of Patients Achieved Remission
Description: The degree of remission of proteinuria obtained (complete or partial) The rate of decline of renal function measured by the Modification of Diet in Renal Disease equation for glomerular filtration rate.
Time Frame: 6-12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tacrolimus | Tacrolimus and Mycophenolate Mofetil
Number analyzed (Participants) | 20 | 20
Participants | 16 | 19

ADVERSE EVENTS:
Time Frame: 9.5 years
Arm/Group | Tacrolimus | Tacrolimus and Mycophenolate Mofetil
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 7/20 | 3/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tacrolimus (N=20) | Tacrolimus and Mycophenolate Mofetil (N=20)
diarrhoe and vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Haemorrhoidectomy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Cholestatic jaundice (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2008-06-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT00843856/Prot_SAP_000.pdf